CLINICAL TRIAL: NCT05611450
Title: Developing and Testing a Mobile Health Application of Disease Self-Management in Non-Small Cell Lung Cancer Patients During Targeted Therapy: A Mixed-Methods Study
Brief Title: Mobile Health Application of Disease Self-Management in Non-Small Cell Lung Cancer Patients During Targeted Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Kang Hua Chen, Associate Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 202100777B0
Record Dates: First submitted 2022-11-02; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: disease self-management; mobile application; target therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine care (Placebo Comparator)
  Interventions: Other: disease self-management application
- lung cancer self-management (Experimental)
  Interventions: Other: disease self-management application

INTERVENTIONS:
Other: disease self-management application — The mHealth application provide disease self-management knowledge and skills and also has the functions of level of skin toxicity warning, uploading photos of skin toxicity, and interacting with healthcare professionals.

SUMMARY:
The study's purpose is to understand the self-management needs of patients with NSCLC receiving targeted therapy, develop a disease self- management application (mHealth Application), and explore the effect of mHealth application on the self-efficacy and health status of patients receiving targeted therapy for NSCLC.

This study adopts a two-group (pre-and-post-test) design experiment. This study is being conducted over a period of 3 years and is divided in two stages. This study enrolled patients with NSCLC in the outpatient clinic and ward of the Division of Chest Medicine in a northern medical center as the research participants. Stage 1 develop a disease self-management application and understands participants' needs by qualitative study. The participants are a purposive sample of 15-20 patients. Data discontinued when theme saturation is achieved. Stage 2 adopted convenient sampling to enroll 108 patients (54 in the experimental group and 54 in the control group) to evaluate the effectiveness of the disease self-management application. After participant's consent was obtained, this study performed the pre-test and randomized the participants. The experimental group received both routine care and the disease self-management App, while the control group received routine care and part of application. This study collected data before the patients received targeted therapy and in months 1, 3, 6, and 9 after treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

* ≧20 years of age
* diagnosed with advanced NSCLC
* were epidermal growth factor, anaplastic lymphoma kinase...inhibitor-naive

Exclusion Criteria:

* had received other anti-cancer therapy
* were difficulty with verbal expression or cognitive dysfunction

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-11-22 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
European Organization for Research and Treatment of Cancer 30-item core quality of life questionnaire | change from baseline at 1 month
  assessing participants' quality of life
European Organization for Research and Treatment of Cancer 30-item core quality of life questionnaire | change from baseline at 3 month
  assessing participants' quality of life
European Organization for Research and Treatment of Cancer 30-item core quality of life questionnaire | change from baseline at 6 month
  assessing participants' quality of life
European Organization for Research and Treatment of Cancer 30-item core quality of life questionnaire | change from baseline at 9 month
  assessing participants' quality of life
NCI-CTCAE (ver 5.0) guideline | change from baseline at 1 month
  assessing participants' skin toxicity grade
NCI-CTCAE (ver 5.0) guideline | change from baseline at 3 month
  assessing participants' skin toxicity grade
NCI-CTCAE (ver 5.0) guideline | change from baseline at 6 month
  assessing participants' skin toxicity grade
NCI-CTCAE (ver 5.0) guideline | change from baseline at 9 month
  assessing participants' skin toxicity grade

SECONDARY OUTCOMES:
knowledge and skills with disease self-management questionnaire | change from baseline at 1 month
  assessing participants' knowledge and skill ability with disease self-management
knowledge and skills with disease self-management questionnaire | change from baseline at 3 month
  assessing participants' knowledge and skill ability with disease self-management
knowledge and skills with disease self-management questionnaire | change from baseline at 6 month
  assessing participants' knowledge and skill ability with disease self-management
knowledge and skills with disease self-management questionnaire | change from baseline at 9 month
  assessing participants' knowledge and skill ability with disease self-management
disease self-efficacy questionnaire | change from baseline at 1 month
  assessing participants' self-efficacy with disease self-management
disease self-efficacy questionnaire | change from baseline at 3 month
  assessing participants' self-efficacy with disease self-management
disease self-efficacy questionnaire | change from baseline at 6 month
  assessing participants' self-efficacy with disease self-management
disease self-efficacy questionnaire | change from baseline at 9 month
  assessing participants' self-efficacy with disease self-management
Hospital Anxiety and Depression Scale | change from baseline at 1 month
  assessing participants' anxiety and depression
Hospital Anxiety and Depression Scale | change from baseline at 3 month
  assessing participants' anxiety and depression
Hospital Anxiety and Depression Scale | change from baseline at 6 month
  assessing participants' anxiety and depression
Hospital Anxiety and Depression Scale | change from baseline at 9 month
  assessing participants' anxiety and depression
Medical Outcomes Study-Social Support Survey | chang from baseline at 1 month
  assessing participants' social support
Medical Outcomes Study-Social Support Survey | chang from baseline at 3 month
  assessing participants' social support
Medical Outcomes Study-Social Support Survey | chang from baseline at 6 month
  assessing participants' social support
Medical Outcomes Study-Social Support Survey | chang from baseline at 9 month
  assessing participants' social support

IPD SHARING:
Plan to Share IPD: No